CLINICAL TRIAL: NCT00274820
Title: A Phase II Trial of Combination Therapy With Thalidomide, Arsenic Trioxide, Dexamethasone, and Ascorbic Acid (TADA) in Patients With Chronic Idiopathic Myelofibrosis or Overlap Myelodysplastic/Myeloproliferative Disorders
Brief Title: Arsenic Trioxide, Ascorbic Acid, Dexamethasone, and Thalidomide in Myelofibrosis/Myeloproliferative Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4Y04
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Ascorbic Acid; Arsenic Trioxide; Dexamethasone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: ascorbic acid — The dose of ascorbic acid will be 1000 mg PO 2-3 hours prior to ATO infusion. The treatment will follow the same schedule as arsenic trioxide.
  Other Names: vitamin C
Drug: arsenic trioxide — Treatment consists of a loading period of five 0.25 mg/kg ATO doses in the first week, followed by maintenance dosing with 0.25 mg/kg ATO twice weekly for 11 weeks. Loading is usually done Monday through Friday of the first treatment week. Maintenance should be started either 72 or 96 hours after the last loading dose. Thereafter, dosing is twice weekly, following an alternating pattern of 72 and 96 hours. For example, maintenance dosing may be done on Mondays and Thursdays, Tuesdays and Fridays, etc. The same pattern should be followed for the entire maintenance dosing period.
  Other Names: Trisenox®; ATO
Drug: dexamethasone — Dexamethasone will be given at a dose of 4mg PO daily for five days every four weeks (i.e., days 1-5, 29-33, 57-61, 84-88, etc.).
Drug: thalidomide — The dose of thalidomide will be 50 mg PO daily starting day 1. The dose will be increased to 100mg PO daily after two weeks if tolerated and only if patients experience < grade 1 thalidomide-attributed toxicity using CTC criteria.
  Other Names: Thalomid®

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Sometimes when chemotherapy is given, it does not stop the growth of cancer cells. The cancer is said to be resistant to chemotherapy. Giving ascorbic acid may reduce drug resistance and allow the cancer cells to be killed. Thalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. Giving arsenic trioxide together with ascorbic acid, dexamethasone, and thalidomide may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving arsenic trioxide together with ascorbic acid, dexamethasone, and thalidomide works in treating patients with chronic idiopathic myelofibrosis or myelodysplastic or myeloproliferative disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy (in terms of response rate) of arsenic trioxide, ascorbic acid, dexamethasone, and thalidomide in patients with chronic idiopathic myelofibrosis or myelodysplastic/myeloproliferative disorders.

Secondary

* Determine the rate of disease progression or progression to acute leukemia in patients treated with this regimen.
* Assess improvement in bone marrow pathology (including degree of fibrosis, percentage of blasts, and resolution of cytogenetic abnormalities) in patients treated with this regimen.
* Determine time to response in patients treated with this regimen.
* Determine the reduction of spleen size in patients treated with this regimen.
* Measure clinical responses and quality of life in subgroups treated with this regimen.
* Determine the safety of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive arsenic trioxide IV over 1-2 hours for 5 days and oral ascorbic acid once daily for 5 days during week 1. Patients then receive arsenic trioxide and ascorbic acid twice a week in weeks 2-12. Patients also receive oral dexamethasone once daily for 5 days in weeks 1, 5, 9, and 12 and oral thalidomide once or twice daily in weeks 1-12. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and after every course.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Chronic idiopathic myelofibrosis or myelodysplastic/myeloproliferative disorders (MDS/MPD), including the following subtypes:

  * Chronic idiopathic myelofibrosis (with extramedullary hematopoiesis)
  * Chronic myelomonocytic leukemia (CMML)
  * Atypical chronic myeloid leukemia
  * MDS/MPD disease, unclassifiable

    * MDS with ≥ 2+ fibrosis present in the bone marrow
    * Patients with MPD must be negative by fluorescent in situ hybridization (FISH) for the BCR/ABL fusion gene

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy of at least 3 months
* Platelet count > 10,000/mm³
* Bilirubin ≤ 2.5 times upper limit of normal (ULN)
* SGOT and SGPT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Potassium ≥ 4.0 mEq/dL (supplemental electrolytes allowed)
* Magnesium > 1.8 mg/dL (supplemental electrolytes allowed)
* Absolute QTc interval < 460 msec

  * Patients who have a QT > 460 after electrolyte repletion and discontinuation of other unessential QT-prolonging drugs will be excluded
* Negative pregnancy test
* Women of childbearing potential must use medically acceptable birth control (two methods of birth control or at least one highly active method and one additional effective method), starting 4 weeks prior to starting thalidomide, all through thalidomide therapy, and for 4 weeks after discontinuing thalidomide
* Male patients with reproductive potential must use a latex condom every time they have sex with a woman from the time that they start taking thalidomide, all through thalidomide therapy, and for 4 weeks after discontinuing thalidomide
* No sperm or blood donation during study treatment
* Must be willing and able to comply with the FDA-mandated System for Thalidomide Educational Prescribing and Safety (S.T.E.P.S™) program
* No other serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the patient at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent
* No preexisting neurotoxicity/neuropathy ≥ grade 2
* Not pregnant or nursing
* No cardiac conduction defects
* No unstable angina
* No myocardial infarction within the past 6 months
* No congestive heart failure of any cause
* No New York Heart Association class II or greater
* No other significant underlying cardiac dysfunction
* No prior malignancy in the 3 years before treatment in this study (other than curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer)
* No sulfa allergy that would interfere with administration of trimethoprim sulfamethoxazole prophylaxis

  * Patients with sulfa allergies who could instead receive pentamidine prophylaxis also will be excluded
  * Patients with sulfa allergies who can instead receive atovaquone may be included

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior investigational or approved therapy for this disease
* No growth factors within 1 week of study enrollment
* No other concurrent cytotoxic drugs or other investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Response rate at 6 months | at 6months of therapy and followed for at least 4 weeks after
  Patients with any improvement in disease status (hematologic improvement or partial remission for patients with higher risk disease) may continue on study until a major response or complete remission occurs. Study visits will occur weekly for the first four weeks, then every four weeks, for each cycle. Laboratory monitoring to assess hematological parameters will occur weekly for the first four weeks, then every four weeks, for each cycle.

SECONDARY OUTCOMES:
Bone marrow response at 6 months | at 6 months
  Bone marrow aspirate / biopsy for morphology and blast count, iron stain and cytogenetics.
Spleen size at 12 weeks | at 12 weeks
  Ultrasound of the spleen
Quality of life | every 12 weeks
  Patients will complete the FACT-An questionnaire every 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkael A. Sekeres, MD, MS, Study Chair — The Cleveland Clinic
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio